CLINICAL TRIAL: NCT02012764
Title: The CCP Study: Coordinated Programme to Prevent Arthritis - Can We Identify Arthritis at a Pre-clinical Stage ?
Acronym: CCP
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Paul Emery, ARUK Professor of Rheumatology, University of Leeds
Other Study IDs: RR06/7674; 06/Q1205/169 (Other: Research Ethics Committee)
Record Dates: First submitted 2013-11-08; First posted 2013-12-16 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Arthritis; Rheumatoid Arthritis
Keywords: Anti-CCP antibody; Inflammatory arthritis; Rheumatoid arthritis; Musculoskeletal symptom
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA sample currently retained as part of a sub-study for a departmental tissue bank.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Musculoskeletal symptoms - Pre diagnosis: Patients presenting with non-specific musculoskeletal complaints at risk of development of RA.

SUMMARY:
This is a 12-month, prospective, observational cohort trial involving Primary Care Trusts (PCTs) wishing to take part in the study and the Early Arthritis Clinic (Anti-CCP sub-clinic) at Chapel Allerton Hospital. The approximate duration of subject participation will be 12 months and the approximate total duration of the study will be 10 years. Patients who have not developed inflammatory arthritis within the 12 month period will have the opportunity to continue follow up within the clinic on an annual basis with additional visits as clinically indicated until the development of IA.

DETAILED DESCRIPTION:
There is accumulating evidence for the need to identify patients with rheumatoid arthritis (RA) early. Damage occurs early and early treatment is effective. Clearly there is a need to improve ways of identifying these patients.

It is recognised that patients with RA often have non-specific musculoskeletal complaints in the months or years prior to development of RA (unpublished observations). Family members of patients with RA are also at greater risk of developing RA.

Given we know that earlier identification of patients enables earlier treatment and this leads to better long-term outcomes, we need a method of identifying patients at the pre-clinical stage of disease.

C-reactive protein (CRP) is an acute phase reactant, produced by the liver, primarily in response to stimulation by interleukin-6 (IL-6). The lower limit of detection of routine CRP is 8mg/dL (or higher), yet the mean CRP in the general population is <2mg/dL11 (as measured by high sensitivity assays). Therefore, patients with early RA may have low-grade inflammation not detected by routine CRP. This has been demonstrated in patients with established disease12, but no studies have been done in early disease. Disease activity variables correlated with increases in highly-sensitive CRP (hs-CRP) and hs-CRP was better than ESR at predicting disease activity and severity12. Interestingly, on retrospective analysis of blood donor serum, increased levels of hs-CRP have been noted in RA patients during the pre-clinical phase, most commonly within the two years prior to symptom onset13. This suggests immunologic changes occur prior to the development of the symptomatic stage and provides an exciting tool for assisting in the diagnosis of very early inflammatory disease

ELIGIBILITY:
Inclusion Criteria:

For the purpose of this study, "musculoskeletal complaint" is defined as any new joint / muscular symptoms, including (but not limited to)

* Rotator cuff tendonitis / subacromial bursitis
* Carpal tunnel syndrome
* Tendonitis e.g. epicondylitis "New" complaint is defined as a symptom in which the patient has not previously reported to their GP.

GP and Musculoskeletal referred patients:

Subject must fulfil all of the following conditions or characteristics in order to be considered for study enrolment or participation:

1. Is age > 18 years
2. Has a new musculoskeletal complaint or has a family member with RA
3. Is capable of understanding and signing an informed consent form

Rheumatology Clinic referred patients:

Subject must fulfil all of the following conditions or characteristics in order to be considered for study enrolment or participation:

1. Is age > 18 years
2. Has a new musculoskeletal complaint
3. Is capable of understanding and signing an informed consent form
4. Has tested CCP Ab positive

Exclusion Criteria:

GP and Musculoskeletal referred patients:

Subjects with any of the following conditions or characteristics will be excluded

1. Patients with clinical synovitis
2. Patient fulfils 1987 ACR Criteria or the 2010 ACR/EULAR criteria for RA
3. For the MRI imaging component, the following exclusions will apply; pacemaker, surgical clips within the head, certain inner ear implants, neuro-electrical stimulators or metal fragments within the eye or head or eGFR < 45 ml/min/1.73 m2. In patients with previous penetrating trauma to the eye, or patients at high risk of previous metal foreign body injury to the eye (e.g. welding), skull x-ray will be performed; these patients may be included in the absence of residual metal fragments on x-ray.

Rheumatology clinic referred patients:

Subjects with any of the following conditions or characteristics will be excluded

1. Patient has tested CCP Ab negative
2. Patient fulfils 1987ACR Criteria or the 2010 ACR/EULAR criteria for RA
3. For the MRI imaging component, the following exclusions will apply; pacemaker, surgical clips within the head, certain inner ear implants, neuro-electrical stimulators or metal fragments within the eye or head or eGFR < 45 ml/min/1.73 m2. In patients with previous penetrating trauma to the eye, or patients at high risk of previous metal foreign body injury to the eye (e.g. welding), skull x-ray will be performed; these patients may be included in the absence of residual metal fragments on x-ray.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are attending GP Practices in the Yorkshire and surrounding regions.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2007-01; Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Anti-CCP Ab (+). | 12 years
  The primary objective of this study is to determine the proportion of community patients with new-onset, non-specific musculoskeletal complaints who are anti-CCP Ab (+).

SECONDARY OUTCOMES:
Anti-CCP positive developing I.A | 1 year
  Secondary objectives in this study include:
  1. The number of anti-CCP positive patients who develop an inflammatory arthritis by 12 months / after 12 months.
  * Defined as symptoms and signs of synovitis.
  * Synovitis is defined as the presence soft tissue swelling and at least 1 of the following 2 criteria; tenderness or decreased range of motion.
Anti-CCP positive developing RA | 1 year
  The number of anti-CCP positive patients who develop RA by 12 months/ after 12 months (defined by 1987 ACR and the 2010 ACR/EULAR criteria).
Presenting complaints | 1 week
  To document the initial presenting complaint of all patients (anti-CCP positive and negative)
Predictors for the development of an IA. | 12 years
  To determine usefulness of hs-CRP in predicting development of an IA in patients with positive anti-CCP Ab.
  To determine usefulness of MRI and HRUS in predicting development of an IA in patients with positive anti-CCP Ab.
First degree familymembers who are anti-CCP Ab (+) | 10 years
  To determine the percentage of people with family members who have RA who are anti-CCP Ab (+)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Emery, Study Chair — University of Leeds
Locations (1):
- Chapel Allerton Hospital : Leeds Institute of Rheumatic and Musculoskeletal Medicine, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Garcia-Montoya L, Kang J, Duquenne L, Di Matteo A, Nam JL, Harnden K, Chowdhury R, Mankia K, Emery P. Factors associated with resolution of ultrasound subclinical synovitis in anti-CCP-positive individuals with musculoskeletal symptoms: a UK prospective cohort study. Lancet Rheumatol. 2024 Feb;6(2):e72-e80. doi: 10.1016/S2665-9913(23)00305-3. PMID 38267105
- [Derived] Garcia-Montoya L, Nam JL, Duquenne L, Villota-Eraso C, Di Matteo A, Hartley C, Mankia K, Emery P. Prioritising referrals of individuals at-risk of RA: guidance based on results of a 10-year national primary care observational study. Arthritis Res Ther. 2022 Jan 18;24(1):26. doi: 10.1186/s13075-022-02717-w. PMID 35042555
- [Derived] Ouboussad L, Hunt L, Hensor EMA, Nam JL, Barnes NA, Emery P, McDermott MF, Buch MH. Profiling microRNAs in individuals at risk of progression to rheumatoid arthritis. Arthritis Res Ther. 2017 Dec 22;19(1):288. doi: 10.1186/s13075-017-1492-9. PMID 29273071
- [Derived] Nam JL, Hensor EM, Hunt L, Conaghan PG, Wakefield RJ, Emery P. Ultrasound findings predict progression to inflammatory arthritis in anti-CCP antibody-positive patients without clinical synovitis. Ann Rheum Dis. 2016 Dec;75(12):2060-2067. doi: 10.1136/annrheumdis-2015-208235. Epub 2016 Jan 22. PMID 26802181
- [Derived] Nam JL, Hunt L, Hensor EM, Emery P. Enriching case selection for imminent RA: the use of anti-CCP antibodies in individuals with new non-specific musculoskeletal symptoms - a cohort study. Ann Rheum Dis. 2016 Aug;75(8):1452-6. doi: 10.1136/annrheumdis-2015-207871. Epub 2015 Sep 22. PMID 26395501
- [Derived] Rakieh C, Nam JL, Hunt L, Hensor EM, Das S, Bissell LA, Villeneuve E, McGonagle D, Hodgson R, Grainger A, Wakefield RJ, Conaghan PG, Emery P. Predicting the development of clinical arthritis in anti-CCP positive individuals with non-specific musculoskeletal symptoms: a prospective observational cohort study. Ann Rheum Dis. 2015 Sep;74(9):1659-66. doi: 10.1136/annrheumdis-2014-205227. Epub 2014 Apr 12. PMID 24728331